CLINICAL TRIAL: NCT01300767
Title: 4 Week Performance Comparison Between 2 Commercially Available Silicone Hydrogel Lenses
Brief Title: Four Week Performance Comparison Between Two Commercially Available Silicone Hydrogel Lenses
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: CIBA VISION (Industry)
Responsible Party: Sponsor
Organization: Alcon Research (Industry)
Allocation: Randomized | Model: Single Group | Masking: Single | Purpose: Treatment
Other Study IDs: P-336-C-019
Record Dates: First submitted 2011-02-18; First posted 2011-02-23 (Estimated); Results first posted 2012-05-09 (Estimated); Last update posted 2012-07-10 (Estimated); Status verified 2012-04

CONDITIONS: Myopia
MeSH Terms: conditions — Myopia

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No

ARMS (2):
- Lotrafilcon B (Experimental): Lotrafilcon B commercially marketed contact lens randomly assigned to one eye, with balafilcon A commercially marketed contact lens in the fellow eye for contralateral wear. Lenses were worn for approximately 5 days or more per week, at least 10 hours per day, for up to 4 weeks in a daily wear (DW) modality.
  Interventions: Device: Lotrafilcon B contact lens (AIR OPTIX® AQUA); Device: Contact lens solution (Clear Care®)
- Balafilcon A (Active Comparator): Balafilcon A commercially marketed contact lens randomly assigned to one eye, with lotrafilcon B commercially marketed contact lens in the fellow eye for contralateral wear. Lenses were worn for approximately 5 days or more per week, at least 10 hours per day, for up to 4 weeks in a daily wear (DW) modality.
  Interventions: Device: Balafilcon A contact lens (PureVision® 2); Device: Contact lens solution (Clear Care®)

INTERVENTIONS:
Device: Lotrafilcon B contact lens (AIR OPTIX® AQUA) — Silicone hydrogel, single vision contact lens worn in one eye in a daily wear modality for approximately 5 days or more per week, at least 10 hours per day, for up to 4 weeks.
  Other Names: AIR OPTIX® AQUA
  Arms: Lotrafilcon B
Device: Balafilcon A contact lens (PureVision® 2) — Silicone hydrogel, single vision contact lens worn in one eye in a daily wear modality for approximately 5 days or more per week, at least 10 hours per day, for up to 4 weeks.
  Other Names: PureVision® 2
  Arms: Balafilcon A
Device: Contact lens solution (Clear Care®) — Hydrogen peroxide-based system used for cleaning, disinfection and overnight storage of the study contact lenses.
  Other Names: Clear Care®

SUMMARY:
The purpose of this study is to compare the performance of two commercially marketed contact lenses when worn for up to 4 weeks in a daily wear modality.

ELIGIBILITY:
Inclusion Criteria:

* Habitual spherical soft contact lens wearer who wears a contact lens brand with a recommended replacement schedule of 2 weeks or greater.
* Have a need for correction in both eyes and be correctable to at least 20/40 distance vision in each eye at the dispense of study lenses.
* Willing and able to wear spherical contact lenses within the available range of powers.
* Wears contact lenses at least 5 days per week and at least 10 hours per day, removing them nightly.
* Other protocol-defined inclusion criteria may apply.

Exclusion Criteria:

* Eye injury or surgery within twelve weeks prior to enrollment.
* Currently enrolled in any clinical trial.
* Any use of medications for which contact lens wear could be contraindicated as determined by the investigator.
* Astigmatism of 1.00D or more.
* Currently wearing contact lenses in a daily disposable modality.
* Currently wearing AIR OPTIX AQUA or PureVision 2 contact lenses
* Currently sleeping overnight in contact lenses on an occasional or extended wear basis.
* Other protocol-defined exclusion criteria may apply.

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 75 (Actual)
Dates: Start 2011-02; Primary Completion 2011-04 (Actual); Study Completion 2011-04 (Actual)

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Participants were recruited from 5 US study centers.
Pre-assignment Details: • One participant was enrolled but not dispensed due to failing inclusion/exclusion criteria. This participant is included in the Actual Enrollment calculation, but not in the Participant Flow or Baseline Characteristics calculations.
Groups:
- Lotrafilcon B /Balafilcon A: Lotrafilcon B commercially marketed contact lens randomly assigned to one eye, with balafilcon A commercially marketed contact lens in the fellow eye for contralateral wear. Lenses were worn in a daily wear (DW) modality for approximately 5 days or more per week, at least 10 hours per day, for up to 4 weeks.
Period: Overall Study
Arm/Group | Lotrafilcon B /Balafilcon A
Started | 74
Completed | 70
Not Completed | 4
Not completed — Discomfort | 2
Not completed — Biomicroscopy | 1
Not completed — Unacceptable fit | 1

BASELINE CHARACTERISTICS:
Arm/Group | Lotrafilcon B /Balafilcon A
Number analyzed (Participants) | 74
Age Continuous [Mean (Standard Deviation); unit: years] | 32.8 (10.1)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 54
  Male | 20

OUTCOME MEASURES:

1. Primary Outcome: Comfort on Insertion
Description: As interpreted and recorded by the participant on a questionnaire as a single, retrospective evaluation of 4 weeks of wear. Comfort on insertion was graded on a 10-point scale, with 1 being poor and 10 being excellent.
Time Frame: 4 weeks
Population: Analysis conducted per protocol, with exclusions due to reasons such as, major protocol deviations as determined by masked review; discontinuations; and/or missing responses.
Measure: Mean (Standard Deviation); unit: Units on a Scale
Groups:
- Lotrafilcon B: Lotrafilcon B commercially marketed contact lens randomly assigned to one eye and worn for up to 4 weeks in a daily wear DW) modality.
- Balafilcon A: Balafilcon A commercially marketed contact lens randomly assigned to one eye and worn for up to 4 weeks in a daily wear (DW) modality.
Arm/Group | Lotrafilcon B | Balafilcon A
Number analyzed (Participants) | 70 | 70
Units on a Scale | 8.3 (1.6) | 7.5 (2.0)

2. Primary Outcome: Comfort During the Day
Description: As interpreted and recorded by the participant on a questionnaire as a single, retrospective evaluation of 4 weeks of wear. Comfort during the day was graded on a 10-point scale, with 1 being poor and 10 being excellent.
Time Frame: 4 weeks
Measure: Mean (Standard Deviation); unit: Units on a Scale
Arm/Group | Lotrafilcon B | Balafilcon A
Number analyzed (Participants) | 70 | 70
Units on a Scale | 7.9 (1.8) | 7.2 (2.0)

3. Primary Outcome: Comfort at End of Day
Description: As interpreted and recorded by the participant on a questionnaire as a single, retrospective evaluation of 4 weeks of wear. Comfort at end of day was graded on a 10-point scale, with 1 being poor and 10 being excellent.
Time Frame: 4 weeks
Measure: Mean (Standard Deviation); unit: Units on a Scale
Arm/Group | Lotrafilcon B | Balafilcon A
Number analyzed (Participants) | 70 | 70
Units on a Scale | 7.1 (2.3) | 6.4 (2.3)

4. Primary Outcome: Overall Comfort
Description: As interpreted and recorded by the participant on a questionnaire as a single, retrospective evaluation of 4 weeks of wear. Overall comfort was graded on a 10-point scale, with 1 being poor and 10 being excellent.
Time Frame: 4 weeks
Measure: Mean (Standard Deviation); unit: Units on a Scale
Arm/Group | Lotrafilcon B | Balafilcon A
Number analyzed (Participants) | 70 | 70
Units on a Scale | 7.7 (1.9) | 6.9 (2.1)

5. Primary Outcome: Daytime Vision
Description: As interpreted and recorded by the participant on a questionnaire as a single, retrospective evaluation of 4 weeks of wear. Daytime vision was graded on a 10-point scale, with 1 being poor and 10 being excellent.
Time Frame: 4 weeks
Measure: Mean (Standard Deviation); unit: Units on a Scale
Arm/Group | Lotrafilcon B | Balafilcon A
Number analyzed (Participants) | 70 | 70
Units on a Scale | 8.7 (1.4) | 8.5 (1.5)

6. Primary Outcome: Low Light Vision
Description: As interpreted and recorded by the participant on a questionnaire as a single, retrospective evaluation of 4 weeks of wear. Low light vision was graded on a 10-point scale, with 1 being poor and 10 being excellent.
Time Frame: 4 weeks
Measure: Mean (Standard Deviation); unit: Units on a Scale
Arm/Group | Lotrafilcon B | Balafilcon A
Number analyzed (Participants) | 70 | 70
Units on a Scale | 8.5 (1.4) | 8.3 (1.6)

7. Primary Outcome: Handling on Insertion
Description: As interpreted and recorded by the participant on a questionnaire as a single, retrospective evaluation of 4 weeks of wear. Handling on insertion was graded on a 10-point scale, with 1 being difficult and 10 being easy.
Time Frame: 4 weeks
Measure: Mean (Standard Deviation); unit: Units on a Scale
Arm/Group | Lotrafilcon B | Balafilcon A
Number analyzed (Participants) | 70 | 69
Units on a Scale | 8.5 (1.8) | 7.5 (2.4)

8. Primary Outcome: Handling at Removal
Description: As interpreted and recorded by the participant on a questionnaire as a single, retrospective evaluation of 4 weeks of wear. Handling at removal was graded on a 10-point scale, with 1 being difficult and 10 being easy.
Time Frame: 4 weeks
Measure: Mean (Standard Deviation); unit: Units on a Scale
Arm/Group | Lotrafilcon B | Balafilcon A
Number analyzed (Participants) | 70 | 69
Units on a Scale | 8.5 (1.8) | 7.9 (2.2)

9. Primary Outcome: Delivers a Healthy, Natural Feeling
Description: As interpreted and recorded by the participant on a questionnaire as a single, retrospective evaluation of 4 weeks of wear. Delivers a healthy, natural feeling was graded on a 10-point scale, with 1 being poor and 10 being excellent.
Time Frame: 4 weeks
Measure: Mean (Standard Deviation); unit: Units on a Scale
Arm/Group | Lotrafilcon B | Balafilcon A
Number analyzed (Participants) | 70 | 70
Units on a Scale | 7.9 (2.0) | 6.8 (2.5)

10. Primary Outcome: Lens Awareness
Description: As interpreted and recorded by the participant on a questionnaire as a single, retrospective evaluation of 4 weeks of wear. Lens awareness was graded on a 10-point scale, with 1 being very aware and 10 being not aware.
Time Frame: 4 weeks
Measure: Mean (Standard Deviation); unit: Units on a Scale
Arm/Group | Lotrafilcon B | Balafilcon A
Number analyzed (Participants) | 70 | 70
Units on a Scale | 7.7 (2.3) | 6.2 (2.8)

11. Primary Outcome: Overall Satisfaction
Description: As interpreted and recorded by the participant on a questionnaire as a single, retrospective evaluation of 4 weeks of wear. Overall satisfaction was graded on a 10-point scale, with 1 being poor and 10 being excellent.
Time Frame: 4 weeks
Measure: Mean (Standard Deviation); unit: Units on a Scale
Arm/Group | Lotrafilcon B | Balafilcon A
Number analyzed (Participants) | 70 | 70
Units on a Scale | 7.8 (2.1) | 6.6 (2.3)

12. Primary Outcome: Purchase Intent
Description: As interpreted and recorded by the participant on a questionnaire as a single, retrospective evaluation of 4 weeks of wear. The participant was asked, "How likely would you be to purchase these lenses?" Purchase intent was graded on a 5-point Likert scale: Definitely would purchase, probably would purchase, may or may not purchase, probably would not purchase, definitely would not purchase. The Top-2-box response (definitely would purchase, probably would purchase) was calculated and reported as a percentage of all responses.
Time Frame: 4 weeks
Measure: Number; unit: Percent likely to purchase
Arm/Group | Lotrafilcon B | Balafilcon A
Number analyzed (Participants) | 70 | 70
Percent likely to purchase | 64.3 | 35.7

ADVERSE EVENTS:
Time Frame: Adverse events were collected for the duration of the trial: 09 FEB 2011 to 07 APR 2011.
Description: This reporting group includes all enrolled and dispensed participants.
Arm/Group | Lotrafilcon B | Balafilcon A
Serious Adverse Events (participants affected / at risk) | 0/74 | 0/74
Other Adverse Events (participants affected / at risk) | 0/74 | 0/74

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
For a period of 10 years, the clinical investigator must hold all trial-related information and documents confidential and must agree to obtain sponsor's written consent before discussing, presenting, publicizing, or otherwise disclosing any preclinical and/or clinical data or impressions from this trial.